CLINICAL TRIAL: NCT06869824
Title: A Randomized, Double-blind, Placebo-controlled Trial of the Efficacy of Minayo Iron-rich Nutritional Gummies on Female Anemia, Skin Condition and Qi-blood Deficiency Syndrome
Brief Title: The Efficacy of Minayo Iron-rich Nutritional Gummies on Female Anemia, Skin Condition and Qi-blood Deficiency Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Agile Groups Network Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25-RD-01-MY-001
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Anemia; Skin Condition; Qi-blood Deficiency Syndrome
Keywords: Minayo; Iron-rich Nutritional Gummies; Serum ferritin; Hemoglobin
MeSH Terms: conditions — Anemia; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minayo Iron-rich Nutritional Gummies (Active Comparator): Minayo Iron-rich Nutritional Gummies, 3g/piece, each piece contains 7mg of iron.
  Main ingredients: Maltitol liquid, isomaltitol, erythritol, gelatin, ferrous gluconate, ferrous fumarate, ferric ammonium citrate, acerola cherry powder, cranberry powder, red beetroot powder, raspberry powder, acai powder, salmon hydrolyzed protein peptides, blood protein polypeptides, albumin peptides, Vitamin B1, Vitamin B2, Vitamin B6, Vitamin C, α-cyclodextrin, purple carrot concentrated juice, grape skin extract, agar, citric acid, DL-malic acid, natural food flavoring, octane, glyceryl caprate, and carnauba wax ..
  Interventions: Dietary Supplement: Minayo Iron-rich Nutritional Gummies
- Common Gummies (Placebo Comparator): common gummies with main ingredient - Maltodextrin, 3g/piece
  Interventions: Dietary Supplement: Common Gummies

INTERVENTIONS:
Dietary Supplement: Minayo Iron-rich Nutritional Gummies — Participants need to eat one piece of the assigned product after meal three times a day, for 4 consecutive weeks.
  Arms: Minayo Iron-rich Nutritional Gummies
Dietary Supplement: Common Gummies — Participants need to eat one piece of the assigned product after meal three times a day, for 4 consecutive weeks.
  Arms: Common Gummies

SUMMARY:
The goal of this randomized, double-blind, placebo controlled study is to learn about the efficacy of Minayo Iron-rich Nutritional Gummies on females who are aged 18-45 and suffer nutritional Anemia, skin condition and Qi-blood deficiency syndrome. The main question it aims to answer is:

- whether the Anemia (measured by serum ferritin level and hemoglobin concentration Level in blood) is improved after the intervention

36 qualified participants will be enrolled and assigned to two equal-size groups with study product (Minayo Iron-rich Nutritional Gummies) and placebo product (common gummies) in one study center in Shanghai. The study will last 4 weeks and three site visits will be made, during which all clinical data will be captured and entered to EDC system for statistical analysis and reporting.

Researchers will find out whether the study product (Minayo Iron-rich Nutritional Gummies) is effective to improve Anemia, skin conditions, and Qi-blood deficiency symptoms by comparing the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, aged 18 to 45;
* 36 young women with mild anemia (hemoglobin value between 90-110 g/l) were recruited based on WHO diagnostic criteria for anemia. 10 of the subjects always have coffee and milk tea more than once per day;
* Participants agree not to take any drugs, supplements, or other dairy products during the trial;
* Participants agree not to take any other medications or supplements containing iron during the trial;
* Antibiotics may be used unless medically required, but the type and dosage and days taken should be recorded;
* Willing to refrain from participating in other interventional clinical studies during the trial period;
* Fully understand the nature, purpose, benefits and possible risks and side effects of the study;
* Willing to obey all test requirements and procedures;
* Sign informed consent form.

Exclusion Criteria:

* Anemia due to organic conditions;
* Subject who is in the treatment of gastrointestinal symptoms;
* Lactose intolerance;
* Subject who is currently presence of other organic diseases affecting intestinal function, such as history of gastrointestinal resection, colon or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, congenital megacolon, scleroderma, anorexia nervosa, etc.;
* Controlling diet, exercising, or taking medications to control weight or affect appetite in the last 3 months;
* Subject who has any of the following medical history or clinical findings that may affect the evaluation of the trial effect: significant gastrointestinal disorders, liver, kidney, endocrine, hematological, respiratory and cardiovascular diseases;
* Abuse alcohol or other drugs, supplement or OTC drugs currently or in the past may cause bowel dysfunction or can affect test result evaluation;
* Frequently use of medications that may affect gastrointestinal function or the immune system according to investigator's judgment;
* Take laxatives or other substances that promote digestion 2 weeks before the trail start;
* Subject who used drugs or supplements of iron agent 10 days before the beginning of the trial;
* Pregnant or lactating women or those planning to become pregnant during the trial;
* PI deems that subjects could not fully cooperate with trial arrangements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female subjects, aged 18 to 45
Enrollment: 36 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-04-13 (Actual)

PRIMARY OUTCOMES:
Change of Serum Ferritin Level | baseline day, end of week 4
  The change of serum ferritin level in blood, ng/mL (12~135ng/mL for healthy female, 27~375ng/mL for healthy male)
Change of Hemoglobin Concentration Level | baseline day, end of week 4
  The change of hemoglobin concentration level in blood, g/L (115-150g/L)

SECONDARY OUTCOMES:
Facial image capturing and analysis | baseline day, end of week 4
  The facial images capturing and analysis by VISIA-CR® imaging system, the degree of facial ruddiness/redness, number of wrinkle lines
Change of hand temperature | baseline day, end of week 4
  The change of hand temperature in celsius degree measured by FLIR E60 thermal imaging camera

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — Raison Biotech Co., Ltd
Locations (1):
- Shanghai Raison CMA Lab, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No